

## Tyumen Cardiology Research Center, Tomsk National Research Medical Center, Russian Academy of Science, Tomsk, Russia

Effect of introducer length on the rate of radial artery occlusion during endovascular coronary procedures: a pilot randomized clinical trial (146)

Statistical Analysis Plan

Statistical processing of the obtained data will carried out using statistical software package (SPSS Inc., version 21.0). Results will be presented as  $M \pm SD$  at normal distribution; the values will be represented by the median with an interquartile range, Me (25%; 75%) at asymmetric distribution. The distribution of quantitative variables will be evaluated using the Kolmogorov-Smirnov criterion. Comparing quantitative variables, the nonparametric Mann-Whitney criterion will be applied. The Fisher criterion will be used to compare qualitative variables. Differences between groups will be considered statistically significant at p<0.05.